CLINICAL TRIAL: NCT06447766
Title: A Clinical-Community Partnership to Promote Food Access and Parental Feeding Practices: A Pilot Feasibility Trial
Brief Title: Pediatric Parental Feeding Video Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1914742-6
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Food Insecurity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Education Videos (Experimental): Receive weekly nutrition education videos about evidence-based parental feeding practices and food assistance programs.
  Interventions: Behavioral: Feeding Families Your Way Program

INTERVENTIONS:
Behavioral: Feeding Families Your Way Program — Feeding Families Your Way is a video-based education program delivered by the University of Rhode Island Supplemental Nutrition Assistance Program - Education (SNAP-Ed).

SUMMARY:
The goal of this clinical trial is to learn about the acceptability and feasibility of nutrition education videos among food-insecure parents and caregivers of young children (under 8 years old).

Participants will:

* Watch short nutrition education videos weekly for 8 weeks.
* Complete demographic and nutrition behavior questionnaires at week 1 and week 8.
* Participate in three motivational interview phone calls with a nutrition educator lasting 20 minutes over the course of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Screen positive for food insecurity at Hasbro Children's Hospital Primary Care Clinic.
* Parent or caregiver of at least one child between 3-8 years old.
* Speak English or Spanish fluently.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Food Security Status | 8 weeks
  Two-item food security screener adapted from Hunger Vital Sign.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No